CLINICAL TRIAL: NCT01946100
Title: A Clinical Pathway for the Treatment of Multifocal Lung Adenocarcinoma Using Genome Sequencing
Brief Title: Treatment of Multifocal Lung Adenocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended prior to completion of enrollment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, MD, PhD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-007569
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lung Neoplasms; Carcinoma Non-small-cell Lung; Adenocarcinoma
Keywords: multifocal; genetic; bronchoalveolar carcinoma; adenocarcinoma in situ; ground glass opacity; next generation sequencing
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multifocal Lung Adenocarcinoma (Other)
  Interventions: Genetic: Multifocal Lung Adenocarcinoma

INTERVENTIONS:
Genetic: Multifocal Lung Adenocarcinoma — Tissue collection at the time of surgery for genetic testing and blood sample for germ line DNA.

SUMMARY:
To gather preliminary safety and outcome data for the multimodality treatment of lung adenocarcinoma in the setting of multifocal BAC.

DETAILED DESCRIPTION:
Lung bronchoalveolar carcinoma (BAC) or adenocarcinoma in situ (AIS) continues to represent a poorly understood clinical entity. A frequent clinical dilemma in lung cancer care is the management of a documented or suspected invasive adenocarcinoma in the setting of multifocal ground glass opacity (GGO) consistent with multifocal AIS. These patients are typically classified as stage IV disease, and treated with palliative chemotherapy. No existing pathologic or molecular test is currently capable of making the distinction between independent primary versus metastatic tumors, a distinction for which substantial treatment impact exists. Many treating physicians suspect that outcomes for this specific patient subgroup are better than norms for stage IV disease, as such patients are frequently node-negative and without distant metastases despite multiple lesions present. To address this issue, we will evaluate a multimodality treatment protocol using aggressive local and targeted systemic therapy for multifocal lung adenocarcinoma, incorporating information from tumor genome sequencing for individualized treatment planning. The results will have significant impact in advancing the biologic understanding and treatment approach for lung adenocarcinoma in the setting of multifocal AIS.

ELIGIBILITY:
* Patient must be > 18 years of age
* Two or more GGO's or solid lesions suspicious for multifocal disease.
* Clinical diagnosis of N0
* No evidence of distant metastases
* No prior intra-thoracic radiation therapy (NOTE: Previous radiotherapy as part of treatment for head and neck, breast, or other non-thoracic cancer is permitted.), previous chemotherapy, or surgical resection for non-small cell lung cancer (NSCLC).
* No other cancer in the past 5 years except early stage prostate cancer, or basal cell of skin.
* PFT's that show patient is capable of tolerating a lung resection.
* Non-pregnant and non-lactating. Women of child-bearing potential must have a negative urine or serum pregnancy test to participate in the study.
* Patient must be able to understand and willing to sign an IRB-approved informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11-06 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Overall survival compared to survival for Stage IV NSCLC on NCCTG trials

SECONDARY OUTCOMES:
Progressive free survival | Every 3 months for 2 years
  Progressive free survival
Treatment Morbidity and Mortality | 2 years
  Treatment Morbidity and Mortality
Post-treatment Pulmonary Function | 2 years
  Post-treatment Pulmonary Function measured by pulmonary function testing (spirometry)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Saddoughi SA, Powell C, Stroh GR, Rajagopalan S, Bartholmai BJ, Boland JM, Aubry MC, Harmsen WS, Blackmon SH, Cassivi SD, Nichols FC, Reisenauer JS, Shen KR, Mansfield AS, Maldonado F, Peikert T, Wigle DA. Long-Term Survival and CANARY-Based Artificial Intelligence for Multifocal Lung Adenocarcinoma. Mayo Clin Proc Digit Health. 2024 Jan 11;2(1):44-52. doi: 10.1016/j.mcpdig.2023.10.006. eCollection 2024 Mar. PMID 40206677